CLINICAL TRIAL: NCT02128828
Title: H020: Single-Arm Open Label, Pilot Study of CCR5/CCR2 Inhibitor Cenicriviroc (CVC) for HIV Associated Neurocognitive Disorder (HAND)
Brief Title: Effect of Cenicriviroc on HIV Neurocognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Cecilia Shikuma, Professor, Dept of Medicine, University of Hawaii
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H020
Record Dates: First submitted 2013-09-04; First posted 2014-05-01 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: AIDS Dementia Complex; HIV-1-Associated Cognitive Motor Complex; Human Immunodeficiency Virus
Keywords: AIDS Dementia Complex; HIV-1-Associated Cognitive Motor Complex; Human Immunodeficiency Virus
MeSH Terms: conditions — AIDS Dementia Complex; Acquired Immunodeficiency Syndrome | interventions — cenicriviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cenicriviroc (Experimental): cenicriviroc 50 mg tablets, number of tablets adjusted for other antiretroviral medications or other drugs, given once daily
  Interventions: Drug: cenicriviroc

INTERVENTIONS:
Drug: cenicriviroc — cenicriviroc given once daily for 24 weeks; number of pills dependent on recommended modifications based on patient's other antiretroviral medications and certain other medications anticipated to interact with cenicriviroc
  Other Names: TBR-652

SUMMARY:
The study hypothesis is that cenicriviroc will improve cognition in HIV infected individuals with cognitive impairment. The investigators will study the effect of cenicriviroc on cognition in 24 subjects over a 24 week period.

DETAILED DESCRIPTION:
HIV-associated neurocognitive disease (HAND), particularly in its milder form, is estimated to occur in greater than 30% of HIV infected individuals in the era of potent antiretroviral therapy. As even mild disease leads to functional consequences with decreased ability to live independently, HAND is of substantial public health concern. HIV-induced immune activation/inflammation of monocytes (MO) may be primarily responsible for the development of HAND.

Cenicriviroc is a combined CCR5 and CCR2 chemokine co-receptor antagonist. The investigators hypothesize that dual CCR5 and CCR2 blockade with the use of CVC will lead to measurable reductions in MO activation and lead to cognitive improvement by decreasing HIV infection of MO and by interrupting the trafficking of such MO into the central nervous system.

The investigators propose a single arm, 24-week trial of CVC in 24 subjects with HIV-1 infection suppressed on ART (plasma HIV RNA < 50 copies/ml) for 1 year or more with mild to moderate cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* 4.2.1.1 Documentation of HIV-1 infection by an FDA approved test at any time prior to study entry
* On ARV medication uninterrupted for > 1 year leading up to the screening period
* Screening plasma HIV RNA < 50 copies/ml within 3 months of entry
* Willingness for males and females of childbearing potential to utilize 2 effective contraception methods (2 separate forms, one of which must be an effective barrier method), be non-heterosexually active or have a an exclusive vasectomized partner from screening throughout the duration of the study treatment and for 30 days following the last dose of study drugs.
* Age 18 to 70 years
* Ability and willingness to provide written informed consent
* Mild to moderate cognitive impairment with global neuropsychological (NP) test (NPZglobal) score of < -0.5 or a neurocognitive abnormality (<-0.5) in at least one cognitive domain known to be typically affected by HIV OR unimpaired
* On antiretroviral (ARV) therapy consisting of nucleoside reverse transcriptase inhibitors, atazanavir with/or without ritonavir, darunavir plus ritonavir, dolutegravir, raltegravir or efavirenz.

Exclusion Criteria:

* Receiving or used a CCR5 antagonist within 6 months of study entry
* Plasma HIV RNA > 100 copies/ml within 6 mo. of screening
* HIV-2
* Chronic hepatitis B (positive hepatitis B surface antigen)
* Chronic hepatitis C (positive hepatitis C antibody), except with proof of viral clearance and normal liver function tests
* Active or chronic liver disease
* Active or inadequately treated tuberculosis infection, or inadequate treatment for a positive purified protein derivative test. Adequate treatment meets current recommendations of the Center for Disease Control, NIH and the HIV Medicine Association of the Infectious Diseases Society of America (IDSA) guidelines or other Center for Disease Control recommendations if patient was treated before the current recommendations or before coinfection with HIV.
* Prior/current diagnosis with other intracellular pathogens (Listeria monocytogenes, Toxoplasma gondii, and Cryptococcus neoformans).
* Uncontrolled seizures
* Current or past malignancies excluding basal cell cancer and Kaposi's sarcoma (skin).
* Immunomodulator, HIV vaccine, any other vaccine, or investigational therapy within 30 days of entry.
* Requirement for acute therapy for AIDS-defining or other serious medical illnesses within 14 days of entry.
* Other chronic illnesses including hematologic, pulmonary, autoimmune diseases and endocrinopathies, except for stable controlled diabetes or cardiovascular disease in the view of the investigator and stable testosterone or thyroid therapy.
* Known hypersensitivity to CVC or its excipients
* Anticipated need for prescription medication not allowed in the study. Unwilling to stop eating grapefruit or using St. John's wort).
* Chronic use of over the counter medications unless approved by Study Investigator
* Hemoglobin < 8.5; Absolute neutrophil count < 1000; Platelet count < 100,000; serum glutamate oxaloacetate and pyruvate transaminase > 2.5x upper limit of normal ; Lipase > 2.0 x upper limit of normal
* Estimated creatinine clearance < 30 mL/min(Cockcroft and Gault 1979)
* Bradycardia, sinus rhythm <50 beats/min (bpm).
* Presence of any condition that would interfere with the absorption, distribution, metabolism, or excretion of the drug
* Current active illicit substance or alcohol use or abuse which, in the judgment of the Investigator, will interfere with the patient's ability to comply with protocol requirements
* Pregnancy or breast-feeding
* History of moderate (Child-Pugh class B) or severe (Child-Pugh C) hepatic impairment
* Patients, who, in the opinion of the Investigator, are unable to comply with the dosing schedule and protocol evaluation or for whom the study may not be advisable
* For MRI substudy [impaired]: Any factor that precludes MRI scan including presence of metal or exposure to metal work (e.g. metal grinder/worker) and claustrophobia
* For MRI substudy [impaired]: Any central nervous system pathology which, in the judgment of the investigator, will interfere with the ability to assess study change in magnetic resonance spectroscopy
* 4.2.2.28 For lumbar puncture substudy: Thrombocytopenia or other bleeding disorders (including ongoing anticoagulant therapy), suspected increased intracranial pressure or spinal epidural abscess, or any other factor which would increase risk of complications following lumbar puncture

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Shikuma, MD, Principal Investigator — University of Hawaii - Hawaii Center for AIDS (HICFA)
Locations (1):
- Clint Spencer Clinic, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cenicriviroc
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cenicriviroc
Number analyzed (Participants) | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [46 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Global Neuropsychological Performance
Description: Raw scores from individual performance on 14 validated neuropsychological tests meant to assess various cognitive domains were converted into standardized z-scores adjusted for age, sex, and education. Z-scores from all tests were aggregated and averaged to determine each subject's Global Neuropsychological Performance Score; NPZ-Global). Z-scores follow a normal distribution with scores < '0' identifying poorer cognition than 'average' and scores > "0" identifying better cognition than average with -1 and +1 represented 1 SD below or higher than average.
Time Frame: baseline, week 24
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cenicriviroc
Number analyzed (Participants) | 17
units on a scale | .24 [-.03 to .46]
Statistical Analysis 1: Comparison: Cenicriviroc; Test type: Superiority; p = 0.0079, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Cenicriviroc
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 9/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cenicriviroc (N=20)
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Loose stools (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No